CLINICAL TRIAL: NCT01224743
Title: Effect of Fruit and Vegetable Concentrates on Endothelial Function in Persons With Metabolic Syndrome: A Randomized, Controlled, Crossover Trial
Brief Title: Effect of Fruit and Vegetable Concentrates on Endothelial Function in Persons With Metabolic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: NSA, LLC (Industry)
Responsible Party: David L. Katz, MD, MPH / Director, Yale-Griffin Prevention Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2004-22
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Gardens; Farms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo capsules are provided by the study sponsor and are identical in appearance to active treatments to ensure blinding.
  Interventions: Dietary Supplement: Placebo
- Blend 2 (Experimental): Blend 2 - combination of Juice Plus+® Orchard (Fruit) and Garden (Vegetable) blends
  Interventions: Dietary Supplement: Blend 2
- Blend 1 (Experimental): Blend 1 - combination of Juice Plus+® Orchard (Fruit), Garden (Vegetable), and Vineyard (Berry) blends
  Interventions: Dietary Supplement: Blend 1

INTERVENTIONS:
Dietary Supplement: Blend 1 — Blend 1 consists of a combination of Juice Plus+® Orchard (Fruit), Garden (Vegetable), and Vineyard (Berry) blends
  Other Names: Juice Plus+® Orchard, Garden, Vineyard
  Arms: Blend 1
Dietary Supplement: Blend 2 — Blend 2 consists of a combination of Juice Plus+® Orchard (Fruit) and Garden (Vegetable) blends
  Other Names: Juice Plus+® Orchard, Garden
  Arms: Blend 2
Dietary Supplement: Placebo — Placebo capsules are provided by the study sponsor and are identical in appearance to active treatments to ensure blinding.
  Arms: Placebo

SUMMARY:
Dehydrated fruit and vegetable concentrates provide an accessible form of phytonutrient supplementation that may offer cardioprotective effects. This study assessed the effects of encapsulated fruit and vegetable juice powder concentrates on endothelial function and cardiac risk markers in subjects in a randomized, double blind, placebo controlled crossover clinical trial with three treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome defined by AHA/NHLBI criteria
* nonsmoker
* not taking any other vitamins or dietary supplements
* able to have blood pressure measured bilaterally at the brachial artery

Exclusion Criteria:

* any unstable medical condition that would limit the ability to participate fully in the trial
* rheumatologic disease requiring regular use of NSAIDs
* preexisting cardiovascular disease
* diagnosed eating disorder
* inability to complete endothelial function assessment.
* use of insulin, glucose sensitizing medication, vasoactive medications (including glucocorticoids, antineoplastic agents, psychoactive agents, or bronchodilators), nutriceuticals, fiber supplements, and tobacco.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 8-weeks
  Endothelial function as flow-mediated dilatation (FMD)

SECONDARY OUTCOMES:
Weight | 8-weeks
  Measured on a calibrated scale
Lipid panel | 8-weeks
  Total cholesterol, TG, HDL, LDL, ratio
Insulin | 8-weeks
  Serum insulin

CONTACTS AND LOCATIONS:
Overall Officials: David L Katz, MD, MPH, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Griffin Hospital, Derby, Connecticut, United States

REFERENCES:
- [Derived] Ali A, Yazaki Y, Njike VY, Ma Y, Katz DL. Effect of fruit and vegetable concentrates on endothelial function in metabolic syndrome: a randomized controlled trial. Nutr J. 2011 Jun 29;10:72. doi: 10.1186/1475-2891-10-72. PMID 21714890